CLINICAL TRIAL: NCT05228171
Title: Use of a Mobile Food Record, Enhanced by a Novel Artificial Intelligence-Based Informatics Framework to Expand Capture of Dietary Intake
Brief Title: Mobile Food Record on Recall Effects
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: MED-2021-30429
Record Dates: First submitted 2022-01-21; First posted 2022-02-08 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-02

CONDITIONS: Healthy
Keywords: Mobile food record; nutrition

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Standard Recall: Standard interviewer-administered 24-hour dietary recall.
- Augmented Recall: Interviewer use of the mCC app for 24-hour dietary recall.
  Interventions: Behavioral: mCC app

INTERVENTIONS:
Behavioral: mCC app — Interviewer use of the mCC app during the 24-hour dietary recall interview.
  Groups: Augmented Recall

SUMMARY:
Human dietary habits remain challenging to measure. Even the "gold-standard" interviewer-administered 24 hour dietary recall has established underreporting issues especially in high-risk populations, such as patients with obesity. Performance of precision nutrition research requires state of the art tools to capture individual dietary patterns. Given the widespread availability of smart phones, mobile-phone based food records present a prime opportunity to capture "in the field" dietary intake. Mobile food records, however, are not yet widely used in nutrition research. Several reasons exist. First, the mobile food record needs to be validated relative to the "gold standard" of dietary intake, the 24-hour dietary recall. Second, many available mobile food records are commercially based, with caveats about data availability and meeting research-quality data security practices (HIPAA compliance).

In response, this study includes using a freely available, research-focused, HIPAA compliant, mobile food record (mCC: my Circadian Clock app) actively used in research studies (including our own ongoing work) to test the hypothesis that a mobile food record can expand capture of dietary intake. The proposed aims include the following: Using a randomized, cross-over design, evaluation of augmenting interviewer-administered 24-hour dietary recalls by a mobile food record (Augmented Recall) results in less energy intake underreporting than a standard (un-augmented) interviewer administered 24-hour dietary recall (Standard Recall).

ELIGIBILITY:
Inclusion Criteria:

* Adults between 18-65 years old
* BMI ≥30 kg/m2
* Without a 4 year (BS/BA) college degree
* Owns a smart phone
* Able to read and speak English

Exclusion Criteria:

• Pregnant or lactating women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy adults
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2022-03-14 (Actual); Primary Completion 2022-07-12 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Caloric intake | 60 days from intervention
  Compare caloric intake assessed by the augmented recall relative to the standardized recall

SECONDARY OUTCOMES:
Energy intake | 24 hours following food intake
  Comparison of the energy intake calculated from the 24 hour interviewer administered dietary recall which is augmented by concurrent use and review of a mobile food record (Augmented Recall) vs the energy intake calculated from standard interviewer administered 24-hour dietary recall (Standard Recall)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Chow, MD, Principal Investigator — UMN
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No